CLINICAL TRIAL: NCT04407676
Title: A Randomised Controlled Trial of Enhanced Informed Consent Compared to Standard Informed Consent To Improve Patient Understanding of Early Phase Oncology Clinical Trials
Brief Title: Improving Informed Consent for Early Phase Anti-Cancer Trials
Acronym: CONSENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR 5165
Record Dates: First submitted 2020-05-21; First posted 2020-05-29 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Solid Neoplasms
Keywords: Drug Development; Informed consent; Clinical Trials

STUDY DESIGN:
Intervention Model Description: Randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients eligible for an investigator initiated trial are given the standard PIS by email, and are also emailed a summary PIS and access to an online set of 10 video educational modules. They are then administered a demographic data collection form, the Quality of Informed Consent Questionnaire Parts A and B, and a user feedback survey form. They then present for their standard of care consent visit.
  Interventions: Other: Summary PIS and Online Video Modules
- Control (Placebo Comparator): Patients eligible for an investigator initiated trial are given the standard PIS by email and are then administered a demographic data collection form, the Quality of Informed Consent Questionnaire Parts A and B, and a user feedback survey form. They will then be emailed and are also emailed a summary PIS and access to an online set of 10 video educational modules. They will then perform the QuIC-A and QuIC-B again. They will then present for their standard of care consent visit.
  Interventions: Other: Summary PIS and Online Video Modules

INTERVENTIONS:
Other: Summary PIS and Online Video Modules — Complex trial information presented in alternative and more accessible formats

SUMMARY:
The purpose of the trial will be to test whether providing both a short summary PIS and a link to a set of online video modules will improve patient understanding (those considering early phase clinical trials) as measured on the Quality of Informed Consent questionnaire (Part A), as compared to a control group who are provided only the normal PIS, and also to assess user acceptability and feasibility of these interventions.

DETAILED DESCRIPTION:
i. General background

Early phase oncology clinical trials are becoming increasingly complex with a rapidly increasing array of investigational agents, combinations of these agents and a variety of trial designs which incorporate the importance of personalised approaches and the hope of fast tracked drug discovery. Informed consent for early phase oncology trials has always been a contentious area, and now it continues to be of relevance for the wider oncology community and the Phase 1 trial community. A 2018 study demonstrated significant gaps in understanding of patients regarding the nature and intent of early phase oncology trials. There has been a longstanding debate in the medical oncology community about the nature of Phase 1 trials and the ethics of allowing vulnerable patients to participate in clinical research where the primary purpose is to establish the safe dose. Opponents of the argument point to the need to understand both sides and that patients need to understand enough to consent, which is not necessarily full comprehension. The fact that this group of patients is hopeful, optimistic and desperate has been well characterized and no doubt plays a role in their ability to process information presented to them by the clinical research team.

ii. Empirical research showing patients misunderstand early phase clinical trials

Multiple studies have shown that advanced cancer patients (ACP) misunderstand the nature and purpose of Phase 1 oncology trials. Most recently, Hlubocky et al. demonstrated through audiotaping clinical encounters between 101 ACPs, and 29 oncologists that ACPs had a poor understanding. Only 26% were able to recall the primary purpose of the trial as safety and only 7% were able to recall that there was a risk of major adverse effects such as organ damage. The study also demonstrated deficiencies in clinician communication, with only 40% of encounters containing a direct statement on the research purpose being to establish safety, toxicity and dosage. In 2010, a similar study of 17 oncologists and 52 patients in the United Kingdom showed that several key areas of information including prognosis were omitted from the clinical encounter.Joffe and colleagues also conducted a survey of trial participants (including phase 1, 2 and 3 clinical trials) and investigators and showed significant deficits in understanding. Furthermore, in a survey of 95 patients on Phase 1 trials, Pentz and colleagues demonstrated that 68.4% of patients had a therapeutic misconception by failing to answer two core questions correctly ("Is the research study mostly intending to help research and gain knowledge or mostly intending to help you as a person?" and "Does the research study or your doctor decide the treatments?"). There was also a misunderstanding of the risk associated with participating in an early phase clinical trial and that they do not correctly grasp the key difference between individualized care and clinical research. There was a correlation between lower education and lower family incomes with therapeutic misconception. Overall there is extensive empirical evidence to suggest that a significant proportion of advanced cancer patients considering early phase oncology clinical trials harbour misconceptions about the nature and design of these trials.

iii. Participant Information Sheets are too long, too complex and fail to meet the information needs of patients

It has long been recognised that Participant Information Sheets (PIS) or Informed Consent Forms (ICF) are highly complex and lengthy across all the phases of oncology clinical trials. In 2007, Beardsley and colleagues showed that PIS were increasing in length and that an objective measure of informed consent (the QuIC-A), understanding decreased as PIS's increased in length. There have been no published studies on the PIS used in Phase 1 studies specifically. However, in the era of combination trials, Bayesian adaptive design, and seamless Phase 1/2 designs, the PIS for Phase 1 trials can be particularly complex. There is regulatory requirement for disclosure and there are certain regulatory requirements but these documents have ultimately become unwieldy, disliked by investigators and anecdotally, not read at all by participants. This further magnifies the issues on therapeutic misconception that were highlighted earlier. We note that the Hastings Center has published a 3 page Phase 1 consent form, but to the best of our knowledge this is not in widespread practice. Overall, in this era of increasingly sophisticated trial design, PIS are becoming lengthier and are becoming less useful as adjuncts to the informed consent process.

iv. Paucity of interventional research to improve understanding

We performed a review of the literature looking at interventions that have been tested to improve participant comprehension of Phase 1 trials which yielded two relevant studies. The first, a simulated teaching intervention to improve clinician confidence by Fallowfield et al. (2012) showed that an intensive 8 hour educational intervention on clinicians involved in early phase trials improved their self-confidence along with patient simulator ratings of understanding(7). Secondly, Kass et al. (2009) randomized 288 participants to receive either a 20 minute educational computer based presentation or a standard pamphlet on clinical trials and showed that they could improve patient understanding of trial purpose from 16% to 34%(8) and also showed that there was no significant differences in likelihood of enrollment. We note that there have been multiple efforts directed towards empowering cancer patients in later phase trials including audiovisual techniques such as multimedia presentations(9), question prompt lists(10), and decision aids (11). Promisingly, sponsors are already taking steps towards improving their information sheets and there are already attempts to incorporate audiovisual materials and electronic assessment of patient understanding.

v. Justification for CONSENT

CONSENT will be a randomised controlled trial examining the effect of both a short, jargon-free, plain language participant information sheet and a suite of online educational videos, on participants considering consenting to an investigator initiated trial within the Drug Development Unit. Early phase trials have dramatically changed over the last decade and there have been no interventional studies published in this area in this time and consequently this is a significant area of unmet need for both patients and investigators. This trial will use a validated measure of informed consent (Quality of Informed Consent - Part A) and powered to test a statistical hypothesis, and will also examine the acceptability of the two interventions for patients. While the trial will employ a randomised design, it will ensure all participants are provided access to the enhanced consent materials prior to their actual consent visit to ensure fairness. This trial will be conducted in compliance with the protocol, standard operating procedures, policies, local R&D management guidance, Good Clinical Practice including the UK Policy Framework for Health and Social Care.

Research Governance Framework 2005 (2nd edition)

2. Rationale

Given the ethical imperative to ensure patients understand the nature and conduct of clinical trials, the clearly documented lack of understanding in the literature, we propose this trial to examine whether a pragmatic and deliverable program of "enhanced" informed consent can impact upon patient objective and subjective understanding. The first part of this enhanced consent will be a summary PIS (example attached in appendix) which contains the absolutely necessary information for patients - we have already conducted a qualitative study of patient focus groups and have asked patients directly their priorities. The top three priorities identified patients were

1. Will this trial work for me?
2. What are the side effects?
3. How often do I have to come? This will consist of an easy to understand flowchart.

The second part of this enhanced consent will be an online link to 10 video modules (transcripts attached in appendix) covering key areas of the consent. During the development process of these educational tools, we performed a qualitative analysis of transcripts of interviews of consultants, study managers, clinical fellows, clinical research nurses and patients of the DDU and identified the key areas that the various stakeholders wished to communicate to patients. We asked about the key areas that need to be communicated, common areas of misunderstanding and preferred ways forward of improving patient understanding.

ELIGIBILITY:
Inclusion criteria

1. For randomised participation, patients must be eligible for an Investigator Initiated Trial (IIT) within the Drug Development Unit

   1. RAFMEK (IRAS 102403, CCR 3808, REC ref: 12/LO/1407)
   2. FRAME (IRAS 225064, CCR 4642, REC ref: 17/LO/1473)
   3. ICE-CAP (IRAS 233461, CCR 4720, REC ref: 18/LO/0059), non GBM cohorts
   4. ACE (IRAS Number 211557, CCR 4500, REC ref: 17/LO/0263)
   5. Other IIT trials as they open, however these trials and accompanying study aids will be added as an amendment to CONSENT

   For participation in non-randomised secondary analysis of GBM patients, patients must be eligible for

   a. ICE-CAP (IRAS 233461, CCR 4720, REC ref: 18/LO/0059), GBM cohorts
2. English is the patient's primary language
3. Written (signed and dated) informed consent and be capable of co-operating with study procedures and questionnaire

Exclusion criteria

1. Pre-existing visual, non-cancer related cognitive impairment, or reading impairment
2. Patients who have already consented to a trial or have prior consent knowledge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2023-03-26 (Estimated)

PRIMARY OUTCOMES:
QuIC-A score (Quality of Informed Consent questionnaire - Part A, Objective) | Through study completion, aiming for 34 patients, expected to reach this in 12 months based on historical recruitment rates
  • To determine the QuIC Part A scores following administration of a standard PIS alone, and compare it to the QuIC Part A score following administration of a standard PIS along with a summary PIS and a suite of online educational videos. Minimum score on QuIC-A is 0, highest is 100, and higher scores indicate a higher degree of objective understanding of clinical trial principles.

SECONDARY OUTCOMES:
QuIC- B score (Quality of Informed Consent questionnaire - Part B, Subjective) | Through study completion, aiming for 34 patients, expected to reach this in 12 months based on historical recruitment rates
  • To determine the QuIC Part B scores following administration of a normal PIS alone, and compare it to the QuIC Part B score following administration of a normal PIS along with a summary PIS and a suite of online educational videos. Minimum score on QuIC-B is 0, highest is 100, and higher scores indicate a higher degree of subjective understanding of clinical trial principles.
Control arm analysis | Through study completion, aiming for 34 patients, expected to reach this in 12 months based on historical recruitment rates
  • To determine the changes in QuIC Part A and Part B scores before and after administration of enhanced consent materials
User feedback | Through study completion, aiming for 34 patients, expected to reach this in 12 months based on historical recruitment rates
  • To confirm the acceptability and utility of the summary PIS and educational videos with a user feedback survey
GBM cohort exploratory analysis | Through study completion, aiming for 15 patients, expected to reach this in 12 months based on historical recruitment rates
  QuIC Part A and Part B scores before and after administration of enhanced consent materials in patients recruited to the GBM cohort in the ICE-CAP study

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Lopez, MRCP PhD, Principal Investigator — The Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hlubocky FJ, Kass NE, Roter D, Larson S, Wroblewski KE, Sugarman J, Daugherty CK. Investigator Disclosure and Advanced Cancer Patient Understanding of Informed Consent and Prognosis in Phase I Clinical Trials. J Oncol Pract. 2018 Jun;14(6):e357-e367. doi: 10.1200/JOP.18.00028. Epub 2018 May 22. PMID 29787333
- [Background] Miller FG, Joffe S. Phase 1 oncology trials and informed consent. J Med Ethics. 2013 Dec;39(12):761-4. doi: 10.1136/medethics-2012-100832. Epub 2012 Nov 17. PMID 23161617
- [Background] Dolly SO, Kalaitzaki E, Puglisi M, Stimpson S, Hanwell J, Fandos SS, Stapleton S, Ansari T, Peckitt C, Kaye S, Lopez J, Yap TA, van der Graaf W, de Bono J, Banerji U. A study of motivations and expectations of patients seen in phase 1 oncology clinics. Cancer. 2016 Nov 15;122(22):3501-3508. doi: 10.1002/cncr.30235. Epub 2016 Sep 26. PMID 27716902
- [Background] Jenkins V, Solis-Trapala I, Langridge C, Catt S, Talbot DC, Fallowfield LJ. What oncologists believe they said and what patients believe they heard: an analysis of phase I trial discussions. J Clin Oncol. 2011 Jan 1;29(1):61-8. doi: 10.1200/JCO.2010.30.0814. Epub 2010 Nov 22. PMID 21098322
- [Background] Joffe S, Cook EF, Cleary PD, Clark JW, Weeks JC. Quality of informed consent in cancer clinical trials: a cross-sectional survey. Lancet. 2001 Nov 24;358(9295):1772-7. doi: 10.1016/S0140-6736(01)06805-2. PMID 11734235
- [Background] Koyfman SA, McCabe MS, Emanuel EJ, Grady C. A consent form template for phase I oncology trials. IRB. 2009 Jul-Aug;31(4):1-8. No abstract available. PMID 19697538
- [Background] Fallowfield LJ, Solis-Trapala I, Jenkins VA. Evaluation of an educational program to improve communication with patients about early-phase trial participation. Oncologist. 2012;17(3):377-83. doi: 10.1634/theoncologist.2011-0271. Epub 2012 Mar 1. PMID 22382459
- [Background] Kass NE, Sugarman J, Medley AM, Fogarty LA, Taylor HA, Daugherty CK, Emerson MR, Goodman SN, Hlubocky FJ, Hurwitz HI, Carducci M, Goodwin-Landher A. An intervention to improve cancer patients' understanding of early-phase clinical trials. IRB. 2009 May-Jun;31(3):1-10. No abstract available. PMID 19552233
- [Background] Synnot A, Ryan R, Prictor M, Fetherstonhaugh D, Parker B. Audio-visual presentation of information for informed consent for participation in clinical trials. Cochrane Database Syst Rev. 2014 May 9;2014(5):CD003717. doi: 10.1002/14651858.CD003717.pub3. PMID 24809816
- [Background] Tattersall MH, Jefford M, Martin A, Olver I, Thompson JF, Brown RF, Butow PN. Parallel multicentre randomised trial of a clinical trial question prompt list in patients considering participation in phase 3 cancer treatment trials. BMJ Open. 2017 Mar 1;7(3):e012666. doi: 10.1136/bmjopen-2016-012666. PMID 28249847
- [Background] Juraskova I, Butow P, Bonner C, Bell ML, Smith AB, Seccombe M, Boyle F, Reaby L, Cuzick J, Forbes JF. Improving decision making about clinical trial participation - a randomised controlled trial of a decision aid for women considering participation in the IBIS-II breast cancer prevention trial. Br J Cancer. 2014 Jul 8;111(1):1-7. doi: 10.1038/bjc.2014.144. Epub 2014 Jun 3. PMID 24892447
- [Background] Joffe S, Cook EF, Cleary PD, Clark JW, Weeks JC. Quality of informed consent: a new measure of understanding among research subjects. J Natl Cancer Inst. 2001 Jan 17;93(2):139-47. doi: 10.1093/jnci/93.2.139. PMID 11208884
- [Background] Hoffner B, Bauer-Wu S, Hitchcock-Bryan S, Powell M, Wolanski A, Joffe S. "Entering a Clinical Trial: Is it Right for You?": a randomized study of The Clinical Trials Video and its impact on the informed consent process. Cancer. 2012 Apr 1;118(7):1877-83. doi: 10.1002/cncr.26438. Epub 2011 Aug 25. PMID 22009665
- [Background] Spellecy R, Tarima S, Denzen E, Moore H, Abhyankar S, Dawson P, Foley A, Gersten I, Horwitz M, Idossa L, Joffe S, Kamani N, King R, Lazaryan A, Morris L, Horowitz MM, Majhail NS. Easy-to-Read Informed Consent Form for Hematopoietic Cell Transplantation Clinical Trials: Results from the Blood and Marrow Transplant Clinical Trials Network 1205 Study. Biol Blood Marrow Transplant. 2018 Oct;24(10):2145-2151. doi: 10.1016/j.bbmt.2018.04.014. Epub 2018 Apr 18. PMID 29679770
- [Derived] Pal A, Stapleton S, Yap C, Lai-Kwon J, Daly R, Magkos D, Baikady BR, Minchom A, Banerji U, De Bono J, Karikios D, Boyle F, Lopez J. Study protocol for a randomised controlled trial of enhanced informed consent compared to standard informed consent to improve patient understanding of early phase oncology clinical trials (CONSENT). BMJ Open. 2021 Sep 6;11(9):e049217. doi: 10.1136/bmjopen-2021-049217. PMID 34489282